CLINICAL TRIAL: NCT04733222
Title: Effect of Treadmill Slip- and Trip-perturbation Training on Falls Among Community-dwelling Older Adults: A Randomized, Controlled Trial
Brief Title: Effect of Treadmill Perturbation Training on Falls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg Municipality (Other); Aalborg University (Other); Odense University Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jens Eg Nørgaard, PhD-student, Cand.Scient., Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N-20200089
Record Dates: First submitted 2021-01-22; First posted 2021-02-02 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Accidental Fall; Accident Prevention
Keywords: Aged; Aged, 80 and over; Exercise; Perturbation training; Older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: After the pre-training tests, participants will be randomly allocated to either the perturation or control group. To produce groups of similar size a permuted block randomization will be used. Allocation concealment will be maintained using random block sizes (4, 6, or 8) and by the randomization code only being available for non-blinded research staff.
  The perturbation group will undergo three initial training sessions on two days within a week, and a "booster"-session after six months. The active control group will perform treadmill walking at a preferred speed to match the training dose of the perturbations group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perturbation training (Experimental): Participants randomized to the treadmill perturbation training will initially perform three sessions performed within a week followed by a "booster"-session after six months.
  Interventions: Other: Perturbation training
- Treadmill walking (Active Comparator): Participants randomized to the walking group will undergo three initial sessions within a week and a "booster"-session after six months.
  Interventions: Other: Treadmill walking

INTERVENTIONS:
Other: Perturbation training — The treadmill perturbation training will be performed on a computer-controlled treadmill. The perturbation will be induced by fast forward (slip) or backward (trip) accelerations of the treadmill at specific gait cycle timings. The perturbations will be delivered randomly to enhance the unpredictability. A ceiling-mounted body-harness ensures the safety of the participants.
  Participants will be assigned to three initial sessions of treadmill slip- and trip-perturbation training on two days separated by a week and a "booster"-session after six months. On day 1, participants will first undergo a session 1 with 40 slip perturbations and then a session 2 with 40 trip perturbations. On day 2, participants will undergo a session 3 with 20 slip and 20 trip perturbations in random order. The "booster"-session after six months will be similar to session 3 (20 of each perturbation in random order).
  Arms: Perturbation training
Other: Treadmill walking — Participants allocated to the walking group will walk at a self-selected pace on a computer-controlled treadmill for the same amount of time as the treadmill perturbation training participants.
  Arms: Treadmill walking

SUMMARY:
This parallel, randomized, controlled trial aims to quantify the effects of slip- and trip-perturbation training on fall rates collected over 12 months, compared to time-matched treadmill walking, among community-dwelling older adults (≥65 years).

A sample size calculation estimated that 140 older community-dwelling older adults (≥65 years) are needed. Following baseline measures, the recruited participants will randomly be assigned to either the perturbation or the walking group. The participants in the perturbation group will be assigned to four perturbation training sessions. The walking group will perform four treadmill walking matching the exercise time of the perturbation training. Assessment of the primary outcome, fall rates, will be conducted continuously in 12 months from randomization. When a fall is reported in the fall calendar, a telephone interview will be conducted to assess the circumstances and consequences (e.g., fall-related fractures, fall-related hospital admissions) of the falls. Moreover, assessment of physical, cognitive, and social-psychological outcomes will be made at baseline, post-test, six-month, and 12-months reassessment.

DETAILED DESCRIPTION:
Approximately one-third of older adults fall at least once a year, and about 10% of these falls cause serious injuries such as head injuries and fractures. In fact, falls are the most frequent cause of injuries among older adults and often lead to disability, institutionalization, and premature death.

Multiple fall prevention interventions have been examined to reduce the fall rate, and physical exercise has continuously been proven as an effective and cost-effective approach. However, traditional exercise approaches, such as balance and muscle-strengthening training, have only shown a moderate 20-25% decrease in falls and encounters issues such as poor compliance. Recently, task-specific perturbation training using an overground walkway has been shown to produce quick motor adaptations resulting in improved pro- and reactive stability. Additionally, perturbation training delivered on such walkways has decreased both laboratory-induced and real-life falls. However, overground walkways with moveable platforms and trip-board are expensive and immobile; thus, limiting the clinical feasibility.

Contrarily, perturbation training delivered on computer-controlled treadmills may serve as a more implementable substitute. Preliminary studies have shown that treadmill perturbation training produces similar dynamic stability adaptations to overground perturbation training. Furthermore, a single session of treadmill perturbation decreases the rate of laboratory-induced falls, and the ergogenic effects were retained for up to six months. However, the effects of a brief treadmill perturbation training intervention on real-life falls in community-dwelling older adults still vastly unknown.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years old
* Community-dwelling
* Able to walk without a walking aid

Exclusion Criteria:

* Any of the following self-reported conditions: Any orthopedic surgery within the past 12 months, osteoporosis or history of osteoporosis-related fractures (low impact hip, spine, and wrist fracture), or progressive neurological disease (e.g., Parkinson, multiple sclerosis)
* An unstable medical condition that would prevent safe participation
* Severe cognitive impairment (a score <8 in The Short Orientation-Memory-Concentration Test)
* Current participation in another fall prevention trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Fall rate | Continuously for 12 months after the initial three training sessions
  Falls are collected by daily recordings in calendar that is returned to the research group monthly

SECONDARY OUTCOMES:
Proportion of participants with at least one fall | Continuously for 12 months after the initial three training sessions
  Falls are collected by daily recordings in calendar that is returned to the research group monthly
Time to first fall | Continuously for 12 months after the initial three training sessions
  Falls are collected by daily recordings in calendar that is returned to the research group monthly
Fall-related fracture rate | Continuously for 12 months after the initial three training sessions
  When a fall is registered in the fall calendar, a research group member will make a telephone interview to obtain information about the fall's consequences (e.g. fractures). Screening of the participants medical records for radiologically verified fractures will verify this information.
Proportion of participants with at least one fall-related fractures | Continuously for 12 months after the initial three training sessions
  When a fall is registered in the fall calendar, a research group member will make a telephone interview to obtain information about the fall's consequences (e.g. fractures). Screening of the participants medical records for radiologically verified fractures will verify this information.
Number of all-cause fractures | At the 52-week follow-up
  Screening of the participants medical records for radiologically verified fractures.
Number of other fall-related injuries | Continuously for 12 months after the initial three training sessions
  When a fall is registered in the fall calendar, a research group member will make a telephone interview to obtain information about the fall's consequences (e.g. head injuries and bruises).
Fall-related hospital admission rate | Continuously for 12 months after the initial three training sessions
  When a fall is registered in the fall calendar, a research group member will make a telephone interview to obtain information about the fall's consequences (e.g. hospital contacts). Screening of the participant's medical records will verify this information.
Proportion of participants with at least one hospital admission | Continuously for 12 months after the initial three training sessions
  When a fall is registered in the fall calendar, a research group member will make a telephone interview to obtain information about the fall's consequences (e.g. hospital contacts). Screening of the participant's medical records will verify this information.
Number of all-cause hospital admissions | At the 52-week follow-up
  Screening of the participant's medical records
Laboratory-induced falls | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  Falls after slips and trips induced on the treadmill. A fall is determined based on video recordings. A fall is defined as unambiguous support by the safety harness after the perturbation.
Gait kinematics to perturbations | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  Gait kinematics collected before, during and after a slip- and trip-perturbation measured by heel contacts
Single-task gait | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  8-meter walking timed by handheld stopwatch.
Dual-task gait | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  8-meter walking timed by handheld stopwatch under dual-task condition (serial subtraction of threes from a random three digit number).
Single-task static balance | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  30-seconds static balance measures on a Wii balance board.
Dual-task static balance | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  30-seconds static balance measures on a Wii balance board under dual-task conditions (verbal fluency of grocery store items).
Choice stepping reaction time | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  Choice stepping reactions test on a Wii balance board
Lower extremity physical performance | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  The Short Physical Performance Battery
Health-related quality of life | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  The EuroQoL EQ-5D-5L, Danish version
Fear of Falling | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  The Short Falls Efficacy Scale International, Danish version
Executive function | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  The trail making task Part A and B
Frailty | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  The Tilburg Frailty Indicator
Adverse events | Week 0 (Pre-training; before the first training), week 1 (Post-training; after the third training session), week 26 (26-week follow-up; before the fourth training session), and week 52 (52-week follow-up)
  Patient-reported events such as muscle soreness, discomfort, pain, or injuries

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eg Nørgaard, MSc, Principal Investigator — Aalborg University Hospital and Aalborg University
Locations (1):
- Aalborg Municipality, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norgaard JE, Andersen S, Ryg J, Andreasen J, Oliveira ASC, Stevenson AJT, Danielsen MBB, Jorgensen MG. Perturbation-based balance training of older adults and effects on physiological, cognitive and sociopsychological factors: a secondary analysis from a randomised controlled trial with 12-month follow-up. BMJ Open. 2024 Aug 7;14(8):e080550. doi: 10.1136/bmjopen-2023-080550. PMID 39117404
- [Derived] Norgaard JE, Andersen S, Ryg J, Stevenson AJT, Andreasen J, Oliveira AS, Danielsen MB, Jorgensen MG. Effect of Treadmill Perturbation-Based Balance Training on Fall Rates in Community-Dwelling Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e238422. doi: 10.1001/jamanetworkopen.2023.8422. PMID 37079305
- [Derived] Norgaard JE, Andersen S, Ryg J, Stevenson AJT, Andreasen J, Danielsen MB, Oliveira ASC, Jorgensen MG. Effects of treadmill slip and trip perturbation-based balance training on falls in community-dwelling older adults (STABILITY): study protocol for a randomised controlled trial. BMJ Open. 2022 Feb 7;12(2):e052492. doi: 10.1136/bmjopen-2021-052492. PMID 35131823

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT04733222/Prot_SAP_000.pdf